CLINICAL TRIAL: NCT06057168
Title: Performance of Elucirem (Gadopiclenol) in Dynamic Susceptibility Contrast Magnetic Resonance Imaging (DSC-MRI) Perfusion of Brain Gliomas Phase IIIb Clinical Trial
Brief Title: Performance of Elucirem in DSC-MRI Perfusion of Brain Gliomas
Acronym: GDX-44-016
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GDX-44-016
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor, Primary; Brain Tumor, Recurrent
MeSH Terms: conditions — Brain Neoplasms | interventions — gadopiclenol; gadoterate meglumine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elucirem (Experimental): Patient underwent a DSC-MRI perfusion using Elucirem.
  Interventions: Drug: Elucirem
- Dotarem (Active Comparator): Patient underwent a DSC-MRI perfusion using Dotarem.
  Interventions: Drug: Dotarem

INTERVENTIONS:
Drug: Elucirem — Intravenous administration
  Other Names: gadopiclenol
  Arms: Elucirem
Drug: Dotarem — Intravenous administration
  Other Names: gadoterate meglumine; gadoteric acid
  Arms: Dotarem

SUMMARY:
This trial aimed to study the performance of Elucirem (gadopiclenol) in Dynamic Susceptibility Contrast Magnetic Resonance Imaging (DSC-MRI) perfusion of brain gliomas.

DETAILED DESCRIPTION:
The trial was designed as a prospective, multi-center, randomized, controlled and parallel group comparison.

This study aimed to enrol 138 patients in Italy, Poland and Hungary.

During the course of the trial, patient underwent a DSC-MRI perfusion using Elucirem or Dotarem. A safety visit was performed 1 day after the MRI visit. Confirmation of tumor grade diagnosis, if available, was collected up to 30 days after visit 2. Primary end point was assessed by independent off-site blinded readers.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adult patient (patient having reached legal majority age).
2. Patient with naive or recurrent primary glial tumor detected at a previous Computed Tomography (CT) or MR imaging, and scheduled for a follow-up contrast-enhanced MRI. Tumor grade (confirmed or highly suspected) should be available in patients' medical records.
3. Patient or, if the patient is unable to provide informed consent, the patient's legally acceptable representative and/or impartial witness, having read the information and having provided patient's consent to participate in writing by dating and signing the informed consent prior to any trial related procedure being conducted.
4. Patient affiliated to national health insurance according to local regulatory requirements.

Exclusion Criteria:

1. Patient with known contra-indication(s) to the use or with known sensitivity to one of the products under investigation or to other Gadolinium-Based Contrast Agents (GBCA) (such as hypersensitivity, post-contrast acute kidney injury).
2. Patient presenting with any contraindication to MRI examinations.
3. Post treatment patient presenting with pseudo-progression instead of tumor recurrency.
4. Patient presenting with severe renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m² assessed within 1 week prior to contrast agent injection.
5. Patient having received any contrast agent (for MRI or CT) within 3 days prior to IMP administration or scheduled to receive any contrast agent within 24 hours after IMP administration.
6. Pregnant female patient (a female patient of childbearing potential or with amenorrhea for less than 12 months must have a negative pregnancy test within 1 day prior to trial MRI and must be using medically approved contraception method until the last trial visit).
7. Patient having received any investigational medicinal product within 7 days prior to trial entry or scheduled to receive any investigational treatment in the course of the trial.
8. Patient previously randomized in this trial.
9. Patient with anticipated, current or past condition (medical, psychological, social or geographical) that would compromise the patient's safety or her/his ability to participate in the trial.
10. Patient unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits and/or unlikelihood of completing the trial.
11. Patient related to the investigator or any other trial staff or relative directly involved in the trial conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frantz Hebert, Study Director — Guerbet
Locations (11):
- Hungary (4):
  - Országos Idegtudományi Intézet - Neuroonkológiai és Intracraniá, Budapest
  - Semmelweis Egyetem - Neurologiai Klinika, Budapest
  - Debreceni Egyetem, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Italy (4):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Ospedale San Raffaele- Neuroradiologia, Milan
  - IRCCS C.Mondino, Istituto Neurologico Nazionale, Fondazione, Pavia
  - Policlinico Universitario Agostino Gemelli, Roma
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Szpital Specjalistyczny im.L.Rydygiera, Krakow
  - Independent Public Teaching Hospital no 1 Department of Interventional Radiology and Diagnostic Imaging, Lublin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 141 patients were screened in 10 centers from three countries: 76 from four centers in Hungary, 48 from four centers in Italy and 17 from two centers in Poland.
Pre-assignment Details: Out of the 141 screened patients, 3 patients were screen failed. Therefore, 138 patients were randomized in the trial with 69 in each arm. Out of them, 2 patients prematurely discontinued the study before the injection of contrast agent. The remaining 136 patients underwent MRI examination with injection of IMP: 67 with Elucirem and 69 with Dotarem. A total of 124 patients were included in the per-protocol primary analysis: 60 with Elucirem and 64 with Dotarem.
Groups:
- Elucirem: Patient underwent a DSC-MRI perfusion using Elucirem (gadopiclenol) at 0.05 mmol/kg
  Elucirem: Intravenous administration
- Dotarem: Patient underwent a DSC-MRI perfusion using Dotarem (gadoterate meglumine) at 0.1 mmol/kg
  Dotarem: Intravenous administration
Period: Overall Study
Arm/Group | Elucirem | Dotarem
Started | 69 (69 patients were randomized in the Elucirem group.) | 69 (69 patients were randomized in the Dotarem group.)
Completed | 67 | 69
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline description for safety population (patients received an injection of contrast agent): A total of 136 patients including 67 patients who received an injection of Elucirem and 69 patients who received an injection of Dotarem.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elucirem | Dotarem | Total
Number analyzed (Participants) | 67 | 69 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (14.23) | 54.6 (14.71) | 54.8 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 44 | 39 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 67 | 68 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Quality of Cerebral Blood Volume (CBV) Map of Dynamic Susceptibility Contrast MRI (DSC-MRI) Perfusion
Description: Diagnostic quality of the CBV map obtained from DSC-MRI perfusion for each patient was assessed by the two off-site blinded readers using the following scale (poor, fair, good or excellent) and by a consensus in case of discordance between the two readers. The proportion of patients with "excellent" or "good" diagnostic quality images of Elucirem group was compared to that of Dotarem group. 124 patients (60 with Elucirem and 64 with Dotarem) who had diagnostic CBV map and without major protocol deviation were included in the per-protocol primary analysis.
Time Frame: From beginning to end of procedure for DSC-MRI perfusion using Elucirem or Dotarem
Population: Per-protocol analysis included 124 patients (60 with Elucirem and 64 with Dotarem) with diagnostic CBV map and without protocol major deviation evaluated by two independent off-site readers.
Measure: Count of Participants; unit: Participants
Arm/Group | Elucirem | Dotarem
Number analyzed (Participants) | 60 | 64
Participants | 58 | 63
Statistical Analysis 1: Comparison: Elucirem vs Dotarem; Test type: Non-Inferiority — Non-inferiority was assessed by calculating the difference in proportion of patients presenting with images of excellent or good diagnostic quality between Elucirem and Dotarem groups, and by constructing a two-sided 95% confidence Interval (CI) around this difference. If the lower bound of the two-sided 95% CI was above the pre-stated margin of non-inferiority (-12%), Elucirem was declared non-inferior to Dotarem.The Wald statistical test with a continuity correction was used for CI; Construction of a two-sided 95% CI around the difference in proportion of patients with images of excellent or good diagnostic quality CBV map; two-sided 95% confidence Interval (CI) = -0.018, 95% CI 2-sided [-0.089 to 0.053]

ADVERSE EVENTS:
Time Frame: From the beginning of patient's participation in the trial (Informed Consent Form signature) until the end of the participation (1 day after IMP administration for the patients without biopsy or surgery done, maximum 30 days after IMP administration for the patients with biopsy or surgery done).
Description: AEs occurring during or after IMP administration until the end of the participation (maximum 30 days) for safety population.
  Safety population: the patients who received an IMP of the study (67 patients received an injection of Elucirem group and 69 patients received an injection of Dotarem).
Arm/Group | Elucirem | Dotarem
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/69
Other Adverse Events (participants affected / at risk) | 3/67 | 2/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elucirem (N=67) | Dotarem (N=69)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incorrect dose administered by device (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT06057168/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT06057168/SAP_001.pdf